CLINICAL TRIAL: NCT02911935
Title: Azithromycin to Prevent Wheezing Following Severe RSV Bronchiolitis-II
Acronym: APW-RSV-II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Avraham Beigelman, Associate Professor of Pediatrics, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201603018
Record Dates: First submitted 2016-09-18; First posted 2016-09-22 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Respiratory Syncytial Virus, Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral azithromycin (Active Comparator): Oral Azithromycin
  Interventions: Drug: Oral azithromycin
- Placebo (Placebo Comparator): Oral Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral azithromycin — Oral azithromycin 10mg/kg/day for 7 days; then oral azithromycin 5mg/kg/day for 7 additional days
  Other Names: Azithromycin suspension
  Arms: Oral azithromycin
Drug: Placebo — Placebo suspension
  Arms: Placebo

SUMMARY:
The main objective of the APW-RSV II clinical trial is to evaluate if the addition of azithromycin to routine bronchiolitis care, among infants hospitalized with RSV bronchiolitis, reduces the occurrence of recurrent wheeze during the preschool years.

DETAILED DESCRIPTION:
The APW-RSV II clinical trial is a double blind, placebo-controlled, parallel-group, randomized trial, including otherwise healthy 188 participants, ages 1-18 months, who are hospitalized due to RSV bronchiolitis. The study includes active treatment phase with azithromycin or placebo for 2 weeks, and an observational phase for up to 48 months.

The main objective of the APW-RSV II clinical trial is to evaluate if the addition of azithromycin to routine bronchiolitis care, among infants hospitalized with RSV bronchiolitis, reduces the occurrence of recurrent wheeze (RW) during the preschool years.

Study participants will be enrolled during 3 consecutive RSV seasons beginning in Fall 2016. Study participants will be randomized to receive PO azithromycin 10 mg/kg/day for 7 days followed by 5mg/kg/day for additional 7 days, or matched placebo. The primary clinical outcome is the time to the occurrence of a third episode of wheezing. The duration of follow up is 18-48 months, which is determined based on the year in which the participants is recruited: first year recruits will be followed for up to 48 months, while the 3rd year recruits will be followed for at least 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age: 1-18 months.
* Hospitalization for the first episode of RSV bronchiolitis.
* Confirmed RSV infection by positive nasal swab results (PCR assay and/or direct antigen detection).
* At least two of the following symptoms/signs of bronchiolitis: respiratory rate greater than 40 breaths/minute; cough; wheezing; audible rales, crackles, and/or rhonchi; paradoxical chest movements (retractions)28.
* Duration of respiratory symptoms from onset of symptoms of the current illness to admission is 120 hours (5 days) or less.
* Randomization can be performed within 168 hours (7 days) from onset of symptoms.
* Willingness to provide informed consent by the child's parent or guardian.

Exclusion Criteria:

* Prematurity (gestational age < 36 weeks).
* Presence or history of other significant disease (CNS, lung, cardiac, renal, GI, hepatic disease, hematologic, endocrine or immune disease). Children with atopic dermatitis and/or food allergy will not be excluded from the study.
* Clinically significant gastroesophageal reflux currently treated with a daily anti-reflux medication (anti- H2 or PPI).
* The child has significant developmental delay/failure to thrive, defined as weight < 3% for age and gender.
* History of previous (before the current episode) wheeze or previous (before the current episode) treatment with albuterol.
* History of previous treatment with corticosteroid (systemic or inhaled) for respiratory issues.
* Treatment (past or present) with montelukast.
* Treatment with any macrolide antibiotic (azithromycin, clarithromycin or erythromycin) over the past 4 weeks or current treatment with any macrolide antibiotic. Current or prior treatment with non-macrolide antibiotic is not an exclusion criterion.
* Chronic treatment with any daily medication other than vitamins or nutritional supplements. Although routine vitamin D supplement (400 IU per day) is not an exclusion criterion, high dose vitamin D supplements are not allowed.
* Participation in another clinical trial.
* Participant requires invasive mechanical ventilation due to RSV bronchiolitis.
* Evidence that the family may be unreliable or non-adherent, or has definitive plans to move from the clinical center area before trial completion.
* Contraindication of use of azithromycin or any other macrolide antibiotics such as history of allergic reaction (or other adverse reaction) to these antibiotics.
* Diagnosis of asthma.
* Treatment with other medication that may cause QT interval prolongation.

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Beigelman, MD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Department of Pediatrics, Washington University School of Medicine; and St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to study documents, including the study protocol with any amendments and blank case report forms.
  Upon reasonable request, these data will be provided by Dr. Charles Goss, the study statistician. email: cwgoss@wustl.edu
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: A month after publication
Access Criteria: See above

REFERENCES:
- [Derived] Beigelman A, Goss CW, Wang J, Srinivasan M, Boomer J, Zhou Y, Bram S, Casper TJ, Coverstone AM, Kanchongkittiphon W, Kuklinski C, Storch GA, Schechtman KB, Castro M, Bacharier LB. Azithromycin therapy in infants hospitalized for respiratory syncytial virus bronchiolitis: Airway matrix metalloproteinase-9 levels and subsequent recurrent wheeze. Ann Allergy Asthma Immunol. 2024 May;132(5):623-629. doi: 10.1016/j.anai.2024.01.001. Epub 2024 Jan 17. PMID 38237675
- [Derived] Beigelman A, Srinivasan M, Goss CW, Wang J, Zhou Y, True K, Ahrens E, Burgdorf D, Haslam MD, Boomer J, Bram S, Burnham CD, Casper TJ, Coverstone AM, Kanchongkittiphon W, Kuklinski C, Storch GA, Wallace MA, Yin-DeClue H, Castro M, Schechtman KB, Bacharier LB. Azithromycin to Prevent Recurrent Wheeze Following Severe Respiratory Syncytial Virus Bronchiolitis. NEJM Evid. 2022 Apr;1(4):10.1056/evidoa2100069. doi: 10.1056/evidoa2100069. Epub 2022 Feb 27. PMID 37621674

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: Participants received Azithromycin 10 mg/kg/d orally for 7 days and 5 mg/kg/d orally for additional 7 days
- Placebo: Participants received Azithromycin placebo orally daily for 14 days
Period: Overall Study
Arm/Group | Azithromycin | Placebo
Started | 101 | 99
Completed | 96 | 92
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Azithromycin: Participants orally received Azithromycin 10 mg/kg/d for 7 days and 5 mg/kg/d for additional 7 days
- Placebo: Participants orally received Azithromycin placebo daily for 14 days
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 3.9 [2.3 to 7.2] | 2.8 [1.7 to 6.6] | 3.3 [2 to 6.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 44 | 91
  Male | 54 | 55 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One participant in Placebo arm refused to provide race/ethnicity information
  Participants
    Race and ethnicity: number analyzed (Participants) | 101 | 98 | 199
    Race and ethnicity: African American | 19 | 21 | 40
    Race and ethnicity: Caucasian | 72 | 72 | 144
    Race and ethnicity: More than one race | 10 | 5 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 101 | 99 | 200
Birth weight [Mean (Standard Deviation); unit: kg] | 3.3 (0.5) | 3.4 (0.5) | 3.3 (0.5)
Birth by cesarean section [Count of Participants; unit: Participants] | 29 | 28 | 57
Gestational age at birth [Mean (Standard Deviation); unit: weeks] | 38.9 (1.2) | 38.8 (1.2) | 38.8 (1.2)
Maternal smoking during pregnancy [Count of Participants; unit: Participants] | 19 | 13 | 32
History of breast feeding [Count of Participants; unit: Participants] | 75 | 80 | 155
History of eczema [Count of Participants; unit: Participants] | 16 | 13 | 29
Food allergy diagnosis [Count of Participants; unit: Participants] | 3 | 5 | 8
Parental history of asthma [Count of Participants; unit: Participants] | 33 | 39 | 72
Parental history of other atopic diseases [Count of Participants; unit: Participants] | 60 | 69 | 129
Pet exposure [Count of Participants; unit: Participants] | 59 | 71 | 130
Tobacco smoke exposure [Count of Participants; unit: Participants] | 40 | 26 | 66
Duration of hospital stay [Median (Inter-Quartile Range); unit: hours] — Population: Two patients with missing values were excluded from the analysis population.
  hours
    number analyzed (Participants) | 101 | 97 | 198
    (all) | 51 [33 to 89] | 56 [39 to 77] | 52 [35 to 85]
Duration of oxygen requirement, if required [Median (Inter-Quartile Range); unit: hours] — Population: The analysis population only included infants were supplemented with oxygen if they had oxygen saturation of less than 90% on room air.
  hours
    number analyzed (Participants) | 57 | 57 | 114
    (all) | 46 [26 to 70] | 48 [18 to 62] | 47 [25 to 68]
Lowest oxygen saturation on room air [Mean (Standard Deviation); unit: percentage of oxygen saturation] — Population: Three patients with missing values were excluded from the analysis population.
  percentage of oxygen saturation
    number analyzed (Participants) | 101 | 96 | 197
    (all) | 90.6 (4.4) | 90.7 (5.2) | 90.7 (4.8)
Need for BiPAP ventilation [Count of Participants; unit: Participants] — Population: Two patients with missing values were excluded from the analysis population.
  Participants
    number analyzed (Participants) | 101 | 97 | 198
    (all) | 8 | 5 | 13
Bronchiolitis severity score [Mean (Standard Deviation); unit: Scores on a scale] — Bronchiolitis severity score is the total score of 4 categories including Respiratory rate, Flaring or Retracting, Lowest Oxygen Saturation, and Wheezing. Each category is scored separately and then summed up to get the total score. The score for each category ranges from 0 to 3 with higher numbers indicating worse disease. The total score range from 0-12 with higher numbers indicating worse disease.
  Scores on a scale | 5.3 (1.8) | 5.2 (1.8) | 5.2 (1.8)
Other nonstudy antibiotic (nonmacrolide) use [Count of Participants; unit: Participants] | 30 | 28 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced the Occurrence of a Third Episode of Post-RSV Wheezing (Recurrent Wheeze)
Description: Episodes of wheezing were captured at each of the study telephone interviews and clinic visits using the question, "Has your child's chest sounded wheezy or whistling (with and without a cold)?". A new wheezing episode was defined if at least 7 days without wheezing had been reported since the previous episode.
Time Frame: Follow up duration of 18-48 months
Population: A total of 188 participants (96 in the azithromycin group and 92 in the placebo group) had at least one follow-up visit were included in the final primary outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 96 | 92
Participants | 45 | 33
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; The primary analysis tested the statistical null hypothesis of equal recurrent wheeze rates between the azithromycin and placebo groups; Test type: Superiority; p = 0.08, Log Rank — unadjusted P-value. The threshold for statistical significance was p = 0.05; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.95 to 2.34]
Statistical Analysis 2: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.11, Regression, Cox — p-value is adjusted for race, parental history of asthma, ever exposed to smoke and ever exposed to pets. The threshold for statistical significance was p = 0.05; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.92 to 2.29]

2. Secondary Outcome: Number of Participants Who Had Physician Asthma Diagnosis
Description: Physician asthma diagnosis were captured at each of the study telephone interviews and clinic visits using the question, "Has the doctor told you that your child has asthma?".
Time Frame: Follow up duration of 18-48 months
Population: A total of 188 participants (96 in the azithromycin group and 92 in the placebo group) had at least one follow-up visit were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 96 | 92
Participants | 15 | 8
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.12, Log Rank — Unadjusted. The threshold for statistical significance was p = 0.05; Hazard Ratio (HR) = 1.95, 95% CI 2-sided [0.83 to 4.61]

3. Secondary Outcome: Annualized Number of Days With Respiratory Symptoms (Wheezing, Cough, or Shortness of Breath)
Description: The number of days with respiratory symptoms were captured during clinic visits and by telephone interviews every other month using two questions, "Does your child have coughing, wheezing, shortness of breath or chest tightness during the daytime?", "If yes, estimate the number of days". We used a negative binomial regression analysis with an offset term to adjust for duration of follow-up to get the annualized rate estimate.
Time Frame: Follow up duration of 18-48 months
Population: A total of 188 participants (96 in the azithromycin group and 92 in the placebo group) had at least one follow-up visit were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: days per year
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 96 | 92
days per year | 26.2 [21 to 32.8] | 22.2 [17.7 to 27.9]
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.31, Negative Binomial Regression Analysis — Unadjusted. The threshold for statistical significance was p = 0.05; Rate Ratio = 1.18, 95% CI 2-sided [0.86 to 1.62]

4. Secondary Outcome: Annualized Number of Days With Albuterol Use
Description: The number of days with albuterol use were captured during clinic visits and by telephone interviews every other month using two questions, "Has your child taken Albuterol (also known as Ventolin, Pro-air, Proventil)?" and "please estimate # of days your child had albuterol treatments since the last visit". We used a negative binomial regression analysis with an offset term to adjust for duration of follow-up to get the annualized rate estimate.
Time Frame: Follow up duration of 18-48 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: days per year
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 96 | 92
days per year | 4 [2.4 to 6.6] | 3.3 [2 to 5.4]
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.57, Negative Binomial Regression Analysis — Unadjusted. The threshold for statistical significance was p = 0.05; Rate Ratio = 1.22, 95% CI 2-sided [0.6 to 2.48]

5. Secondary Outcome: Annualized Number of Oral Corticosteroid Courses
Description: The number of oral corticosteroid courses were captured during clinic visits and by telephone interviews every other month using two questions, "Has your child taken Oral steroids (Prednisone, Prednisolone, Orapred, Dexamethasone)?" and "how many separate courses of steroids has your child had since the last visit?". We used a negative binomial regression analysis with an offset term to adjust for duration of follow-up to get the annualized rate estimate.
Time Frame: Follow up duration of 18-48 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: courses per year
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 96 | 92
courses per year | 0.23 [0.15 to 0.35] | 0.17 [0.1 to 0.27]
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.38, Negative Binomial Regression Analysis — unadjusted P-value. The threshold for statistical significance was p = 0.05; Rate Ratio = 1.34, 95% CI 2-sided [0.70 to 2.57]

6. Secondary Outcome: Annualized Number of Antibiotic Courses
Description: The number of antibiotic courses were captured during clinic visits and by telephone interviews every other month using two questions, "Has your child taken any antibiotics?" and "How many separate prescriptions has your child taken of an antibiotic(s)?". We used a negative binomial regression analysis with an offset term to adjust for duration of follow-up to get the annualized rate estimate.
Time Frame: Follow up duration of 18-48 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: courses per year
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 96 | 92
courses per year | 1.2 [0.95 to 1.4] | 1.3 [1 to 1.5]
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.56, Negative Binomial Regression Analysis — Unadjusted. The threshold for statistical significance was p = 0.05; Rate Ratio = 0.92, 95% CI 2-sided [0.7 to 1.22]

7. Secondary Outcome: Number of Participants Who Experienced Serious Adverse Events
Description: Serious Adverse Event were captured during clinic visits and by telephone interviews every other month using designed SAE form.
Time Frame: Follow up duration of 18-48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 101 | 99
Participants | 15 | 16

ADVERSE EVENTS:
Time Frame: Follow up duration of 18-48 months
Groups:
- Azithromycin: Participants orally received azithromycin 10mg/kg/day for 7 days; then oral azithromycin 5mg/kg/day for 7 additional days
- Placebo: Participants orally received placebo daily for 14 days.
Arm/Group | Azithromycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/99
Serious Adverse Events (participants affected / at risk) | 15/101 | 16/99
Other Adverse Events (participants affected / at risk) | 73/101 | 72/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=101) | Placebo (N=99)
Accidental drug ingestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ED visit for gastroenteritis (General disorders) | 0 (0) | 1 (1)
High Fever (Infections and infestations) | 0 (0) | 2 (2)
Hospitalization for bone fracutre (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalization for respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization for wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (2)
Hospitalized for observation and video EEG (Nervous system disorders) | 0 (0) | 1 (1)
Preseptal Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory failure/distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Scheduled surgery for bilateral myringotomy with tube insertion and bilateral Adenotonsillectomy (General disorders) | 0 (0) | 1 (1)
Transferred to PICU during respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hospitalization with hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalized after bronchoscopy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalized for a UTI and fever (Infections and infestations) | 0 (0) | 1 (1)
Hospitalized for dehydration (General disorders) | 0 (0) | 1 (1)
Hospitalized for observation following bronchoscopy, BAL and EGD with biopsies (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalized for planned right open pyeloplasty and observation (General disorders) | 1 (1) | 0 (0)
Hospitalized with respiratory infection (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (4)
Hospitalized with bloody diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hospitalized with questionable seizurelike activity (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalized with pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hospitalized for asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=101) | Placebo (N=99)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5)
Abnormal Neutrophil Count (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Abnormal platelet count (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Acute Otitis Media (Infections and infestations) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1) | 1 (1)
Loose stool (Gastrointestinal disorders) | 3 (3) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Blocked tear duct (Eye disorders) | 1 (1) | 0 (0)
Blood in urine (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Decreased Neutrophil count (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 30 (31) | 21 (21)
Ear infection (Infections and infestations) | 14 (14) | 14 (16)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Fussy (Nervous system disorders) | 0 (0) | 1 (1)
Pink eye (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (General disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 6 (7)
Severe obstructive sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Strep infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 33 (33) | 22 (23)
Vomiting (Gastrointestinal disorders) | 10 (10) | 7 (7)

LIMITATIONS AND CAVEATS:
1. Our ultimate goal was to examine an asthma prevention strategy. However, the primary outcome was defined as recurrent wheeze during 2-4 years of follow-up. This was previously done in other studies in this field.
2. The study primary outcome measure was wheeze assessed by the parents, which has a relatively low correlation with wheeze assessed by physicians. However, a systematic bias is unlikely as both groups were evaluated by the same method

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT02911935/Prot_SAP_000.pdf